CLINICAL TRIAL: NCT01103076
Title: Effects of High Cut-off Hemodialysis on Central Memory CD4+ T Cells and Regulatory T Cells in Patients With End-stage Kidney Disease
Brief Title: Effects of High Cut-off (HCO) Hemodialysis on Central Memory CD4+ T and Treg Cells in Patients With End-stage Kidney Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier du Centre du Valais (Other)
Collaborators: Research Unit CHCVs Hôpital de Sion Switzerland (Unknown); Immunology ICHV Sion Switzerland (Unknown); University of Lausanne Hospitals (Other)
Responsible Party: Pascal Meier MD, CHCVs Hôpital de Sion
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HighCO Hemo study; HCO study (Other: SwissMedic)
Record Dates: First submitted 2010-04-13; First posted 2010-04-14 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2010-03

CONDITIONS: End-stage Kidney Disease; CD4 T Cells; Central Memory T Cells; Regulatory T Cells; Uremic Toxins
Keywords: Immune dysfunction; Hemodialysis; HBV; Vaccination; Immune response
MeSH Terms: conditions — Kidney Failure, Chronic; Immune System Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polyamide 210 H (Active Comparator): Chronic HD patients will be treated in random order with either polyamide or HCO membranes (Polyflux 210 H or HCO 1100) for one month (12 HD sessions) before the crossover.
  Interventions: Device: Polyamide HD membrane
- HCO 1100 (Experimental): Chronic HD patients will be treated in random order with either polyamide or HCO membranes (Polyflux 210 H or HCO 1100) for one month (12 HD sessions) before the crossover.
  Interventions: Device: Polyamide HD membrane

INTERVENTIONS:
Device: Polyamide HD membrane — Single use polyamide membrane

SUMMARY:
In this study, the investigators will evaluate whether CD4+ TCM producing effector cytokines can be distinguished on the basis of their expression of the IL-7 receptor alpha-chain (CD127). Using CD154 production as a marker of Ag-specific CD4+ T cells, the investigators will also test the hypothesis that the phenotype and function of TCM are influenced by the type of Ag they recognize. TCM specific for two cleared protein Ag, tetanus toxoïd (TT) and hepatitis B surface (HBs), inducing an early stage of CD4+ T cell differentiation will be compared to TCM specific for cytomegalovirus (CMV), a persistent virus inducing an advanced stage of CD4+ T cell differentiation.

The primary endpoint is to demonstrate in uremic patients who will begin chronic HD and in patients already chronically hemodialyzed any improvement in CD4+ T cell function ex vivo and in vitro. These analyzes will focus on memory T-cell subsets (i.e. Th17 and Tregs population) using HCO membranes or polyamide dialyzers.

The secondary endpoint is a clinical one, namely, to show any improvement in T cell response to HB and TT vaccination (blood antibody titers).

DETAILED DESCRIPTION:
Chronic hemodialysis (HD) has been associated with changes not only in T cell immunity but also in lipid profile. Apart from their immune function, circulating T cells may participate actively in atherogenesis, and treatments that aim to reduce T cell activation and apoptosis in patients with ESRD reduce the risk for development of cardiovascular disease.

Evidence exists that HD patients are exposed to enhanced oxidative stress that is initiated by the generation of oxygen free radicals, mainly in tissue and probably in the circulation. The most potent O2-generating proteins are oxidatively modified lipoproteins, mainly oxidized (oxLDL). OxLDL have been shown to trigger apoptosis of endothelial cells, macrophages, and lymphocytes. However, the pathophysiological relevance of oxLDL-induced CD4+ T cell apoptosis in HD patients remains uncertain.

Previous findings including ours have suggested that in chronic HD patients, a significantly high percentage of activated CD4+ T cells ultimately do not proliferate but become apoptotic. The induction of activated CD4+ T cell apoptosis from HD patients was dependent on Fas/FasL expression, which leads to a cell contact form of circulating CD4+ T cell self-injury. Furthermore, the investigators showed that activated CD4+ T cells from these patients fail to respond adequately to exogenous IL-2. This is due to the downmodulation of surface IL-2 receptor (IL-2R) beta and gamma subunit expression, impaired IL-2 signal transduction in CD4+ T cells, and/or increased serum levels of soluble IL-2R (sIL-2R). Moreover, in vivo sensitization to IL-2 or low synthesis of endogenous IL-2, themselves potentially may lead to enhanced sensitivity to T cell apoptosis. Decreased proliferative capacity of CD69+/CD4+ T cells that were from individuals with normal renal function and incubated with serum from chronic HD patients and its restoration by normal serum strongly suggest that mediators that are induced by HD affect transduction mechanisms in the IL-2/IL-2R pathway. Finally, IL-2 seems to inhibit the apoptotic process at many stages by interacting with various proteins. Therefore, the investigators postulated that, in HD patients, oxidative stress that is induced by oxLDL may increase CD4+ T cell sensitivity to Fas-mediated apoptosis, in part as a consequence of an HD patient's specific dysregulation of IL-2 expression. To test this hypothesis, the investigators assessed the role of Fas and IL-2 in mediating the oxLDL-induced CD4+ T cell dysfunction in patients with ESRD.

Recently, Meier et al. have shown that HD patients exhibited a reduction in the number of peripheral Tregs, which showed a reduced suppressor function. Considering the oxLDL effects, the relative percentage of Tregs of the total CD4 population was significantly reduced by incubation with oxLDL compared with a nonsignificant depleting effect on CD4+/CD25- T cells. The authors suggest that oxLDL have a specific role on Tregs. More interestingly, Tregs from HD patients exhibited early cell-cycle arrest and became apoptotic. These phenomena were the consequence of the oxLDL-inhibited proteasome proteolytic activity of p27Kip1 and Bax proteins, both of which accumulated in PHA-stimulated Tregs in vitro. Thus, plasma oxLDL in uremic patients might be the trigger of Tregs cycle arrest and apoptosis through proteasome alteration. Furthermore, they found that both uremic serum from HD patients and oxLDL triggered a time- and concentration-dependent down-regulatory effect on the expression of FOXP3. This means that circulating Tregs in HD patients, in addition to being reduced in number, also expressed low levels of FOXP3 per cell, and thus failed to suppress the proliferation of effector cells.

In our study, the investigators want to use gene and protein expression profiling and functional assays of human (ESKD patients on chronic HD or naive uremic patients not yet on HD) CD4+ TCM to identify the mechanisms underlying their maintenance or dysfunction. Our results will provide a molecular basis for the capacity of CD4+ TCM to resist apoptosis and to persist in a stable manner in the host, thereby conferring long-term protective immunity against reinfection. To test this hypothesis, it will be important to determine whether TCM producing cytokines represent a distinct subset of memory cells expressing a specific differentiation phenotype. To the other part the investigators will analyse the role played by Tregs in uremic patients using a new membrane, namely HCO 1100.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESKD (CKD stage 5D according to K/DOQI guidelines) regularly treated by bicarbonate HD 3 times a week for at least 4 h at a blood flow rate of 300 ml/min will be included

Exclusion Criteria:

* Only non-smokers will be enrolled in the study
* Patients with recent (< 3 mo) major trauma, surgery, myocardial infarction, coronary revascularization (coronary angioplasty or bypass surgery), or stroke will be excluded from the study
* Diabetes mellitus
* The presence of an acute or chronic inflammatory process, infection
* Malnutrition (determined by Subjective Global Nutritional Assessment)
* The use of immunosuppressive drugs or evidence of malignancy
* Pregnant women, women who are breast feeding or are of child-bearing potential and not using adequate contraceptive precautions are excluded
* A pregnancy test will be performed in female patients before the inclusion
* Except for aspirin and statin, those patients taking anti-inflammatory medications in the prior 4 weeks will be excluded.
* All patients have to be negative for circulating hepatitis B antigen, hepatitis C antibody (Ab) and HIV
* They will have no active liver disease
* No patient will be nephrectomized
* Arterial blood pH will be between 7.38 and 7.42
* No patient will receive a blood transfusion in the 6 mo before the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-12 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
HCO 1100 membrane effect on T CM and Tregs in patients with ESKD chronically hemodialzed | 12 HD sessions
  The primary endpoint is to demonstrate in uremic patients who will begin chronic HD and in patients already chronically hemodilyzed any improvement in CD4+ T cell function ex vivo and in vitro. These analyzes will focus on memory T-cell subsets (i.e. Th17 and Tregs population) using HCO membranes or polyamide dialyzers.

SECONDARY OUTCOMES:
Immunogenicity of the HB-AS04 vaccine in patients dialyzed with HCO 1100 or polyamide membranes | 12 months study
  The secondary endpoint is a clinical one, namely, to show any improvement in T cell response to HB and TT vaccination (blood antibody titers).

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Meier, MD, Principal Investigator — Nephrology service CHCVs Hôpital de Sion/Switzerland
Locations (1):
- Hôpital de Sion CHCVs, Sion, Valais, Switzerland

REFERENCES:
- [Background] Meier P, Golshayan D, Blanc E, Pascual M, Burnier M. Oxidized LDL modulates apoptosis of regulatory T cells in patients with ESRD. J Am Soc Nephrol. 2009 Jun;20(6):1368-84. doi: 10.1681/ASN.2008070734. Epub 2009 Apr 30. PMID 19406979 (Retraction: PMID 24459234 J Am Soc Nephrol. 2014 Mar;25(3):645)
- [Background] Meier P, Spertini F, Blanc E, Burnier M. Oxidized low-density lipoproteins activate CD4+ T cell apoptosis in patients with end-stage renal disease through Fas engagement. J Am Soc Nephrol. 2007 Jan;18(1):331-42. doi: 10.1681/ASN.2006050514. Epub 2006 Dec 20. PMID 17182885 (Retraction: PMID 24459234 J Am Soc Nephrol. 2014 Mar;25(3):645)
- See also: Centre Hospitalier Universitaire Vaudois — http://www.chuv.ch
- See also: Université de Lausanne — http://www.unil.ch